CLINICAL TRIAL: NCT06330688
Title: Prospective Evaluation of Ultrasound-guided Percutaneous Cholecystostomy With the Trocar Technique
Status: Recruiting | Type: Observational
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Stavros Spiliopoulos, Associate Professor of Diagnostic and Interventional Radiology, Attikon Hospital
Other Study IDs: ΕΒΔ 53/25.01.2024
Record Dates: First submitted 2024-02-22; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Cholecystitis, Acute; Cholecystitis
Keywords: cholecystostomy; percutaneous; trocar; ultrasound; guided; technique; Seldinger; transhepatic; transperitoneal; subcostal; intercostal; technical; success; complications
MeSH Terms: conditions — Cholecystitis, Acute; Cholecystitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: percutaneous cholecystostomy — PC is a minimally invasive, nonsurgical, image-guided intervention that aims to drain and decompress the gallbladder by placing a pigtail catheter through the abdominal wall into the gallbladder lumen.

SUMMARY:
The purpose of this study is to further evaluate and investigate the safety and efficacy of ultrasound (US)-guided percutaneous cholecystostomy (PC) with the trocar technique by the patient's bedside.

DETAILED DESCRIPTION:
This clinical study will include patients who will undergo US-guided PC with the trocar technique. The study will include all cases requiring PC regardless of the underlying cause, while those requiring computed tomography (CT) guidance and those with uncontrolled coagulation disorders will be excluded.

Patient demographics, height, weight, and body mass index (BMI), comorbidities, ASA score, presence or absence of stones, presence or absence of gallbladder perforation at diagnosis, presence or absence of concomitant ascitic effusion, days of preoperative antibiotic treatment, imaging modality used to establish the diagnosis, technical details of the procedure, laboratory values (before and after surgery), and contact information for patient monitoring will be recorded.

The technical success of the method as well as its complications during hospitalization and during a 3-month follow-up period will be calculated. In addition, the anatomical access route during the PC (transhepatic/transperitoneal and intercostal/subcostal), the duration of the operation, the intraoperative and postoperative pain, and the clinical success of the method will be recorded.

After the operation, the patients will be monitored clinically and with laboratory test and, if deemed necessary, US, CT or both imaging will be performed. Before discharge, written instructions will be given regarding the management and care of the catheter.

This study will not burden the hospital financially, as the clinical, laboratory, and imaging tests required for the diagnosis of the underlying etiology that leads to the need to perform the procedure, the technique used to perform the procedure, as well as the monitoring of the patients and the possible complications of the procedure, are part of the hospital's routine.

ELIGIBILITY:
Inclusion Criteria:

* All patients requiring PC, irrespective of the underlying cause and indication, are suitable for inclusion in the study.

Exclusion Criteria:

* Patients are going to be excluded from the study if they are younger than 18 years, if they require PC catheter placement under CT guidance (according to the operator's judgement), or if they suffer from severe uncontrollable coagulopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients requiring PC, irrespective of the underlying cause, comorbidities and indication, and irrespective of patient demographics.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Technical success | Up to 1 hour
  Image verification of correct PC catheter placement within the gallbladder lumen with subsequent bile aspiration at the time of initial catheter placement
Procedure-related complications | Up to 3 months
  Complications attributed to the procedure

SECONDARY OUTCOMES:
duration of the procedure | Up to 1 hour
  The time passed from local anesthesia administration until final pigtail catheter positioning within the gallbladder lumen
intraprocedural and post-procedural pain | Up to 12 hours
  pain experienced during and up to 12 h after the procedure according to the VAS (Visual Analog Scale). The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
clinical success | Up to 72 hours
  The subsidence of signs, symptoms and elevated inflammatory markers up to 72 h after PC (Subsidence of Murphy's sign, pain or tenderness in the right upper quadrant, fever, leukocytosis, elevated C-reactive protein)

CONTACTS AND LOCATIONS:
Locations (1):
- Attikon University Hospital, Chaïdári, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Arkoudis NA, Moschovaki-Zeiger O, Reppas L, Grigoriadis S, Alexopoulou E, Brountzos E, Kelekis N, Spiliopoulos S. Percutaneous cholecystostomy: techniques and applications. Abdom Radiol (NY). 2023 Oct;48(10):3229-3242. doi: 10.1007/s00261-023-03982-2. Epub 2023 Jun 20. PMID 37338588
- [Result] Arkoudis NA, Reppas L, Spiliopoulos S. Image-guided percutaneous cholecystostomy: challenging the norms. Abdom Radiol (NY). 2024 Mar;49(3):939-941. doi: 10.1007/s00261-023-04173-9. Epub 2024 Jan 31. PMID 38294540
- [Result] Arkoudis NA, Moschovaki-Zeiger O, Grigoriadis S, Palialexis K, Reppas L, Filippiadis D, Alexopoulou E, Brountzos E, Kelekis N, Spiliopoulos S. US-guided trocar versus Seldinger technique for percutaneous cholecystostomy (TROSELC II trial). Abdom Radiol (NY). 2023 Jul;48(7):2425-2433. doi: 10.1007/s00261-023-03916-y. Epub 2023 Apr 20. PMID 37081229
- [Result] Reppas L, Arkoudis NA, Spiliopoulos S, Theofanis M, Kitrou PM, Katsanos K, Palialexis K, Filippiadis D, Kelekis A, Karnabatidis D, Kelekis N, Brountzos E. Two-Center Prospective Comparison of the Trocar and Seldinger Techniques for Percutaneous Cholecystostomy. AJR Am J Roentgenol. 2020 Jan;214(1):206-212. doi: 10.2214/AJR.19.21685. Epub 2019 Oct 1. PMID 31573856